CLINICAL TRIAL: NCT02004730
Title: Italian Diffuse/Multivessel Disease ABSORB Prospective Registry Under the Auspices of Società Italiana di Cardiologia Invasive-GISE (IT-DISAPPEARS)
Brief Title: Italian Diffuse/Multivessel Disease ABSORB Prospective Registry: IT-Disappears
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Luca Testa, MD, PhD, I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IT-Disappears
Record Dates: First submitted 2013-11-27; First posted 2013-12-09 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- long single vessel disease (Experimental): ABSORB implantation for long single vessel disease
  Interventions: Device: ABSORB implantation
- multivessel disease ABSORB only (Experimental): multivessel disease treated with ABSORB implantation only
  Interventions: Device: ABSORB implantation
- multivessel disease "hybrid" (Experimental): multivessel disease treated with ABSORB implantation and other devices such as drug eluting stents
  Interventions: Device: ABSORB implantation

INTERVENTIONS:
Device: ABSORB implantation — ABSORB implantation for long (> 24mm) single vessel disease

SUMMARY:
The purpose of this study is to determine whether patients with diffuse or multivessel coronary artery disease may benefit from the percutaneous implantation of the device ABSORB in larger extent with respect to the general population of patients undergoing percutaneous treatment of coronary artery disease.

DETAILED DESCRIPTION:
REGISTRY OBJECTIVE

To investigate the procedural as well as the long-term clinical performance of the ABSORB technology in patients with an indication to percutaneous coronary intervention for:

1. multivessel disease (at least two significant stenosis in 2 different coronary arteries), or
2. long (>24 mm) single vessel disease.

   REGISTRY FLOW AND CLINICAL FOLLOW-UP SCHEDULE

   The Italian National Registry is a prospective multi-center nation-wide registry evaluating the safety and clinical outcomes of the Absorb BVS in daily use in patients with de novo lesions in previously untreated vessels with indication to PCI for multivessel or long single coronary artery disease.

   Indications, however, are per the most recent Absorb IFU.

   Number of Patients to be Registered and Patient Follow-up

   The Italian National Registry will enroll a of 1000 patients in approximately 50 sites throughout the Italian territory where Absorb BVS has regulatory approval and is commercially available.

   Patients will have clinical follow-up by telephone contact or office visits.

   Measures Taken to Avoid and Minimize Bias

   In order to minimize bias in assessing MACE outcomes, these events will be adjudicated by an independent committee.

   Clinical follow-up plan: 30 days, 6 months, 1 year, and then yearly up to 5 years after the index procedure.

   OUTCOMES/ENDPOINTS

   Outcomes are as specified below:

   Primary outcome is set at 1 year: the cumulative hierarchical incidence of major adverse cardiac events (MACE) defined as: cardiac death, non-fatal target vessel myocardial infarction (MI), or clinically driven target lesion revascularization (TLR);

   Secondary endpoints are set at 1 year: All causes mortality, clinically driven TLR, clinically driven target vessel revascularization (TVR), any revascularisation (non TLR, non TVR) and ARC-defined stent thrombosis, at any time point. Any type of angina post procedure measured by means of the Cardio Test, proposed by the ANMCO (Associazione Nazionale Medici Cardiologic Ospedalieri) [21]

   Efficacy parameters: TLR and TVR at 1 year and then yearly up to 5-year follow-up.

   Safety "patient oriented" parameters: at 1 year and then yearly up to 5 years all cause mortality, any myocardial infarction, Stent thrombosis based on the ARC classification, up to 5-year follow-up. Data on dual antiplatelet therapy use will also be collected and analyzed.

   PATIENTS

   Patient Population

   Patients enrolled into this registry will be male and female patients derived from the general interventional cardiology population who satisfy the inclusion and exclusion criteria. The Italian National Registry will enroll 1000 patients in approximately 50 sites throughout the national terrritory.

   Informed Consent

   The Investigator or designee, who has been trained on the protocol, will explain the nature and scope of the registry and inform the patient of the potential risks and benefits of participation, and document consent to treatment with an Absorb BVS device according to standard hospital practice. For this registry the patient must consent to data collection and follow-up visits. All patients (or legally authorized patients' representatives if applicable) must sign, date and time Medical Ethics Committee (MEC) approved informed consent prior to data collection for this registry. Obtaining the consent, provision of a copy to the patient, along with the date and time must be documented in the patient's medical records. The informed consent form must be signed by the investigator. In addition, the signed informed consent must be kept in the patient's medical records.

   Eligibility Criteria

   General Eligibility Criteria

   Assessment for general eligibility criteria is based on medical records of the site and interview with a candidate patient. Patients must meet at least one of the angiographic inclusion criteria to be considered for the registry. If ANY of the exclusion criteria is met, the patient is excluded from the clinical evaluation and cannot be registered.

   Patient Discontinuation

   Once registered, each patient shall remain in the registry until completion of the required follow-up period; however, a patient's participation is voluntary and the patient has the right to withdraw at any time without penalty or loss of benefit. Conceivable reasons for discontinuation may include but not be limited to the following:
   * Patient voluntary withdrawal
   * Patient withdrawal by physician as clinically-indicated
   * Patient lost-to-follow-up: If the patient misses two consecutive scheduled follow up time points, and attempts at contacting the patient are unsuccessful, then the patient is considered lost to follow-up.

   No additional data is needed and will be recorded from patients once withdrawn from the registry. Patients will not be replaced.

   Registry Completion

   An eCRF registry completion form must be completed when:
   * the patient is considered lost-to-follow-up per the above definition or
   * the patient withdraws from the registry or
   * the investigator withdraws the patient from the registry or
   * the patient's follow-up is terminated upon registry follow-up completed

   TREATMENT AND SCHEDULE OF EVENTS

   The treatment strategy will be determined by the investigator. It is required that each enrolling investigator review the most recent Absorb BVS IFU and assess the contraindications, warnings and precaution sections with respect to the risks and benefits for treating potential patients.

   Procedure

   During the procedure, patients will receive appropriate anticoagulation and other therapies according to standard hospital practice. The Absorb BVS will be inspected, prepared, and implanted according to the IFU.

   QCA analysis is recommended pre implantation of the ABSORB, for correct sizing. IVUS, VH-IVUS and OCT techniques are encouraged: these imaging tools will be subject of subgroup analysis.

   Post-procedure (In-hospital)

   Post procedure data will be collected as per eCRF

   Follow-up Antiplatelet Medications

   A minimum of 6 months duration of DAPT is recommended. Specific type of DAPT will be recorded as per eCRF.

   Clinical Follow-up

   Clinical follow-up visits by telephone contact or office visits per the following schedule.
   * 30 days: office visit is encouraged
   * 6 months: office visit is encouraged
   * 1 year, and then yearly up to 5 years after the index procedure: office visit is encouraged.

   Angiographic follow up

   The angiographic follow up will be clinically driven. However, patients undergoing angio follow up and IVUS or OCT follow up will be included in subgroup analysis.

   ADJUDICATION OF EVENTS

   In order to minimize bias in assessing MACE outcomes, these events will be adjudicated by an independent Clinical Event Committee, which will also act as Data Safety and Monitoring Board for the study.

   STATISTICAL ANALYSIS

   Statistical Overview

   The data will be reviewed by a Data Safety and Monitoring Board.

   The Data Safety and Monitoring Board will be also responsible for:
   * Determining whether information collected are sufficient to address the objectives
   * Recommending modifications to the statistical analysis plan to address additional research questions based on review of the data

   Analysis Population

   All patients who are successfully registered will be included in the analysis. A limit of one third of the entire population will be set for the group of Multivessel Disease patients treated with ABSORB and a conventional stent ("hybrid group").

   Sample Size Calculations and Assumptions

   Being this an observational registry aiming at quantifying effect estimates without direct comparisons to literature benchmarks, we relied on confidence interval profiling for sample size justification, without proceeding with formal power analysis. As the main analysis is a pooled analysis of patients with multivessel disease and/or long lesions, an overall and comprehensive analysis is planned as the primary analytical approach. Accordingly, we computed that a target sample of 1000 patients will enable the computation of reasonably precise 95% confidence intervals. Specifically, assuming a 4.2% MACE rate at 1 year (in keeping with ABSORBD EXTEND data), confidence intervals computed with the adjusted Wald method would be 3.1% to 5.6% for a 1000-patient sample (point estimate 42/1000 [4.2%]).

   Given that the registry aims to reflect real-world patients and practice, no provision to limit or restrict patient enrolment depending on the presence of multivessel disease vs long lesions is envisioned.

   Statistical Analyses

   Continuous endpoints will be summarized by presenting the total number of patients, mean, standard deviation, median, minimum, and maximum. Tabulation of categorical parameters will include counts and percentages. The outcomes will be summarized as both a discrete and a continuous variable using the method described above. Survival analysis will be performed with the Kaplan-Meier method. Statistical inference will be based on the computation of 95% confidence intervals using the adjusted Wald method. Additional analyses will involve key subgroups defined according to baseline, lesion, and procedural features, with statistical significance set at the 5% 2-tailed level. Specifically, Student t, Fisher exact, and log-rank tests will be used for such bivariate analyses, whereas multivariable linear regression, logistic regression, and Cox proportional hazard analyses will be used to adjust for confounders. In addition, separate analyses for patients with only multivessel disease, patients with only long lesions, and patients with hybrid revascularization will be performed.

   DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

   The investigator/institution will permit direct access to source data/documents in order for registry-related monitoring, audits, MEC review, and regulatory inspections to be performed.

   As part of the informed consent, the investigator or designee will obtain permission for registry monitors or regulatory authorities to review, in confidence, any records identifying the patients in this registry.

   QUALITY CONTROL AND QUALITY ASSURANCE

   Protocol and Informed Consent Approval The Principal Investigator at each site must confirm and agree with the content of the protocol prior to participation in this registry. Also, the Principal Investigator will obtain written approval of the protocol, informed consent form, and other registry related documents from the MEC. In addition, the investigator will take actions necessary for ongoing registry approval at their site per established procedures of the MEC.

   The investigator will advise the MEC of the progress of this registry on a regular basis until registry completion as required by the MEC.

   The investigator will submit any amendments to the protocol as well as associated informed consent form changes and obtain written MEC approval prior to implementation as required by the MEC.

   Monitoring

   A monitoring plan will be established. Remote monitoring by the CRO and source documents analysis for events throughout the study period by an independent Event Committee, will be conducted to ensure compliance with the protocol and applicable regulatory requirements.

   DATA HANDLING AND RECORD KEEPING

   For the registry duration, the investigator will maintain complete and accurate documentation including but not limited to the following: medical records, registry progress records, laboratory reports, electronic case report forms, signed informed consent forms, device serial numbers for monitoring malfunctions, correspondence with the MEC and registry monitor/Sponsor, SAE reports, and information regarding patient discontinuation or registry completion.

   Source Documentation
   * Medical history/physical condition of the patient before involvement in the registry sufficient to verify protocol entry criteria
   * Dated and signed notes on the day of entry into the registry referencing the sponsor, protocol number, patient ID number and a statement that informed consent was obtained
   * Dated and signed notes from each patient visit
   * Adverse events reported and their resolution including supporting documents such as discharge summaries, catheterization laboratory reports, ECGs, and lab results including documentation of site awareness of SAEs and of investigator device relationship assessment of AEs.
   * Notes regarding Dual Anti Platelet Therapy medications taken during the registry
   * (including start and stop dates)
   * Patient's condition upon completion of or withdrawal from the registry
   * Any other data required to substantiate data entered into the CRF

   Electronic Case Report Form Completion

   Primary data collection based on source-documented hospital and /or clinic chart reviews will be performed clearly and accurately by site personnel trained on the protocol and eCRF completion. eCRF data will be collected for all patients that are registered.

   ETHICAL CONSIDERATION

   Medical Ethics Committee Review Medical Ethics Committee (MEC) approval for the protocol and informed consent form /other written information provided to the patient will be obtained by the Principal Investigator at each investigational site prior to participation in this registry. No changes will be made to the protocol or informed consent form or other written information provided to the patient without appropriate approvals by the MEC.

   Until the registry is completed, the Investigator will advise his/her MEC of the progress of this registry, per MEC requirements.

   Further, any amendments to the protocol as well as associated informed consent form changes will be submitted to the MEC and written approval obtained prior to implementation, according to each institution's MEC requirements.

   APPENDIX I: ABBREVIATIONS AND ACRONYMS

   %DS: percent diameter stenosis AE: adverse event BVS: Bioresorbable Vascular Scaffold CABG: coronary artery bypass graft CE: Conformité Européene (EU) DAPT: Dual Anti Platelet Therapy DES: drug eluting stent eCRF: electronic Case Report Form GCP: Good Clinical Practice IFU: Instructions for Use MACE: major adverse cardiac event MEC: medical ethics committee MI: myocardial infarction PCI: percutaneous coronary intervention PDLLA: Poly-D,L-lactide PLLA: Poly-L-lactide SAE: serious adverse event TLR: target lesion revascularization TVR: target vessel revascularization

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 18 years of age at the time of signing the Informed Consent Form
2. Patient is to be treated for de novo lesions located in previously untreated vessels.
3. Patient must agree to undergo all required follow-up visits and data collection.
4. Patient must have indication to percutaneous coronary intervention for:

   * multivessel disease (at least two significant stenoses in two different segments NOT as a bifurcation lesion; for patients with two vessel disease at least 1 lesion must be >24 mm and must be treated with the BVS; for patients with 3 vessel disease a hybrid approach is acceptable provided that 2 vessels are treated with BVS),

     * long (>24 mm) single vessel disease following:

       1. Stable angina or evidence of myocardial ischemia with stress echocardiography/ myocardial SPECT/exercise test, or
       2. Unstable angina / non ST-elevation myocardial infarction
       3. ST-elevation myocardial infarction with de novo culprit lesion.

Exclusion Criteria:

1. Known intolerance to any of the device components
2. Contraindication to dual antiplatelet therapy (DAPT)
3. Lesion in a saphenous vein graft
4. Lesion to left internal mammary artery
5. Unprotected left main stenosis
6. Woman with childbearing potential
7. Age < 18y/o
8. Concomitant indication to open heart surgery
9. Inability to provide written informed consent
10. Enrolment in another study within 1 month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
the cumulative hierarchical incidence of major adverse cardiac events (MACE) defined as: cardiac death, non-fatal target vessel myocardial infarction (MI), or clinically driven target lesion revascularization (TLR). | 30 days, 6 months, 1 year, and then yearly up to 5 years after the index procedure.

SECONDARY OUTCOMES:
All causes mortality, clinically driven TLR, clinically driven target vessel revascularization (TVR), any revascularisation (non TLR, non TVR) and ARC-defined stent thrombosis, at any time point, any type of angina. | 30 days, 6 months, 1 year, and then yearly up to 5 years after the index procedure.

OTHER OUTCOMES:
Any type of angina post procedure measured by means of the Cardio Test, proposed by the ANMCO (Associazione Nazionale Medici Cardiologic Ospedalieri) | 30 days, 6 months, 1 year, and then yearly up to 5 years after the index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Bedogni, MD, Principal Investigator — Istituto Clinico S. Ambrogio; Anna Sonia Petronio, Prof, Principal Investigator — Univ. of Pisa, Ospedale Cisanello
Locations (2):
- Italy (2):
  - Istituto Clinico S. Ambrogio, Milan
  - Ospedale Cisanello, Pisa

REFERENCES:
- [Derived] De Carlo M, Testa L, Leoncini M, Nicolini E, Varbella F, Cortese B, Ribichini F, Bartorelli AL, Calabria P, Indolfi C, Tomai F, Loi B, Fischietti D, Tarantini G, Bedogni F, Petronio AS. Two-year clinical outcomes of the "Italian diffuse/multivessel disease absorb prospective registry" (IT-DISAPPEARS). Int J Cardiol. 2019 Sep 1;290:21-26. doi: 10.1016/j.ijcard.2019.04.095. Epub 2019 May 3. PMID 31104821
- [Derived] Testa L, Biondi Zoccai G, Tomai F, Ribichini F, Indolfi C, Tamburino C, Bartorelli A, Petronio AS, Bedogni F, De Carlo M. Italian Diffuse/Multivessel Disease ABSORB Prospective Registry (IT-DISAPPEARS). Study design and rationale. J Cardiovasc Med (Hagerstown). 2015 Mar;16(3):253-8. doi: 10.2459/JCM.0000000000000219. PMID 25469734